CLINICAL TRIAL: NCT04370431
Title: A Phase I, Single Center, Randomized, Single-Ascending Dose, Pharmacokinetic and Safety Study (Part A), Bioavailability Comparison Study (Part B) and Food Effect Study (Part C) in Healthy Adult Subjects.
Brief Title: A Study of TTYP01 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Auzone Biological Technology Co., Ltd. (Industry)
Collaborators: TIGERMED AUSTRALIA PTY LIMITED (Unknown); CMAX Clinical Research Pty Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Auzone-01
Record Dates: First submitted 2020-04-18; First posted 2020-05-01 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2021-03

CONDITIONS: Healthy Adult Subjects
MeSH Terms: interventions — Edaravone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- PartA: TTYP01 single ascending doses (Experimental): In Part A: a single-ascending-dose (SAD) escalation study with four consecutive cohorts, single ascending doses of TTYP01 (60, 120, 180 and 240 mg) will be orally administrated.
  Interventions: Drug: TTYP01 single ascending doses
- Part A: Placebo (Placebo Comparator): Placebo control for Part A of the study
  Interventions: Drug: Placebo
- Part B: TTYP01 (oral edaravone) first then IV edaravone (Experimental): Randomized, Open-label, Four-period and Crossover design. A single dose of edaravone in each treatment period. Period 1: 60 mg oral edaravone tablet (TTYP01); Period 2: 30 mg IV edaravone (Radicut® ampoule), Period 3: 120 mg oral edaravone tablet (TTYP01); Period 4: 60 mg IV edaravone (Radicut® bag). Each dose will be spearated by a minimum of 7 days washout period.
  Interventions: Drug: TTYP01, 60 mg; Drug: TTYP01, 120 mg; Drug: Radicut® (ampoule), 30 mg; Drug: Radicut® (bag) , 60 mg
- Part B: IV edaravone first then TTYP01 (oral edaravone) (Experimental): Randomized, Open-label, Four-period and Crossover design. A single dose of edaravone in each treatment period. Period 1: 30 mg IV edaravone (Radicut® ampoule); Period 2: 60 mg oral edaravone tablet (TTYP01); Period 3: 60 mg IV edaravone (Radicut® bag); Period 4: 120 mg oral edaravone tablet (TTYP01). Each dose will be spearated by a minimum of 7 days washout period.
  Interventions: Drug: TTYP01, 60 mg; Drug: TTYP01, 120 mg; Drug: Radicut® (ampoule), 30 mg; Drug: Radicut® (bag) , 60 mg
- Part C: TTYP01: fasted dosing first then fed dosing (Experimental): Randomized, open-Label, Two-period and Crossover design. A fix oral dose of TTYP01 tablet in each treatment period. Period 1: under fasted condition; Period 2: under fed condition. Each dose will be spearated by a minimum of 7 days washout period.
  Interventions: Drug: TTYP01, up to 120 mg
- Part C: TTYP01: fed dosing first then fasted dosing (Experimental): Randomized, open-Label, Two-period and Crossover design. A fix oral dose of TTYP01 tablet in each treatment period. Period 1: under fed condition; Period 2: under fasted condition. Each dose will be spearated by a minimum of 7 days washout period.
  Interventions: Drug: TTYP01, up to 120 mg

INTERVENTIONS:
Drug: TTYP01 single ascending doses — TTYP01 (30 mg edaravone tablet) will be orally administrated at single ascending doses of 60 mg, 120 mg, 180 mg and 240 mg (n=6 per dose)
  Other Names: edaravone tablet
  Arms: PartA: TTYP01 single ascending doses
Drug: Placebo — Placebo control for Part A of the study
  Arms: Part A: Placebo
Drug: TTYP01, 60 mg — TTYP01 oral tablets (30 mg edaravone per tablet)
  Other Names: Edaravone tablet
  Arms: Part B: IV edaravone first then TTYP01 (oral edaravone); Part B: TTYP01 (oral edaravone) first then IV edaravone
Drug: TTYP01, 120 mg — TTYP01 oral tablets (30 mg edaravone per tablet)
  Other Names: Edaravone tablet
  Arms: Part B: IV edaravone first then TTYP01 (oral edaravone); Part B: TTYP01 (oral edaravone) first then IV edaravone
Drug: Radicut® (ampoule), 30 mg — An intravenous dose of edaravone injection, containing 30 mg edaravone in a 20 mL ampoule, will be administered at a dose of 30 mg over 30 minutes
  Other Names: Edaravone injection
  Arms: Part B: IV edaravone first then TTYP01 (oral edaravone); Part B: TTYP01 (oral edaravone) first then IV edaravone
Drug: Radicut® (bag) , 60 mg — An intravenous dose of edaravone injection, containing 30 mg edaravone in a 100 mL injection bag, will be administered at a dose of 60 mg over 60 minutes
  Other Names: Edaravone injection
  Arms: Part B: IV edaravone first then TTYP01 (oral edaravone); Part B: TTYP01 (oral edaravone) first then IV edaravone
Drug: TTYP01, up to 120 mg — TTYP01 oral tablets (30 mg edaravone per tablet). The fixed oral dose level of TTYP01 will depend on the results obtained in Part B of the study (no more than 120 mg)
  Other Names: Edaravone tablet
  Arms: Part C: TTYP01: fasted dosing first then fed dosing; Part C: TTYP01: fed dosing first then fasted dosing

SUMMARY:
This is integrated Phase 1, Single centre, Randomized study will be conducted in 3 parts, each with a specific primary objective:

Part A: To characterise the safety and tolerability of TTYP01 in healthy adult subjects; Part B: To evaluate the bioavailability of TTYP01 tablets in healthy adult subjects; Part C: To characterise the food effect of TTYP01 tablets in healthy adult subjects under the fasted or fed condition.

The secondary objectives of the study are to evaluate the pharmacokinetic (PK) profiles of TTYP01 tablets in healthy adult subjects, and the effects of gender on the PK of TTYP01 tablets in healthy adults. In Part A of the study, a total of 32 healthy adult subjects will be enrolled over four consecutive cohorts (8 per cohort), with participants receiving a single dose of TTYP01 at one of four levels (60, 120, 10 or 240 mg), to assess the PK and safety of TTYP01. In Part B, 16 healthy adults will be randomized into 2 groups, and the comparison of the PK of edaravone (TTYP01 and intravenous (IV) edaravone) will be evaluated using a randomized, open-label, four-period crossover design under fasted conditions. In the first crossover period, subjects will receive a single fixed dose of TTYP01 followed by the alternate IV dose after completion of the washout phase, and in the second crossover period, subjects will receive a higher fixed dose of TTYP01 followed by the alternate IV dose after completion of the washout phase. In Part C, 18 healthy subjects will be enrolled to evaluate the effect of food on the PK of TTYP01 using a randomized, open-label, two-period cross-over design. Participants will be randomized into two groups and administered a fixed dose of TTYP01 on Day 1 (Period 1) under the fed conditions and the second dosing day (Period 2) under the fasted conditions, while the other group being administered a fixed dose of TTYP01 on Day 1 (Period 1) under the fasted conditions and the second dosing day (Period 2) under the fed conditions.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 40, inclusive;
* Non-smokers, ex-smokers and moderate smokers will be included. "A moderate smoker is defined as someone smoking 5 cigarettes or less per day, an ex-smoker is someone who completely stopped smoking for at least 3 months.";
* If female, must be of non-childbearing potential (defined as either surgically sterilized or at least 1 year postmenopausal) or must agree to use a clinically acceptable method of contraception (e.g., oral, intrauterine device [IUD; diaphragm], injectable, transdermal or implantable contraception) or abstinence, for at least 1 month prior to randomization, during the study and 3 month following completion of the study. Females of childbearing potential must have a negative serum human chorionic gonadotropin (hCG) pregnancy test at screening;
* Body Mass Index (BMI) of 18 to 30 kg/m2, inclusive; and a total body weight >50 kg at screening for male subjects, total body weight > 45 kg for female subjects;
* Female subjects of child bearing potential and all male participants who have not had a vasectomy must use effective contraception during the study
* Ability to understand and willingness to sign a written informed consent form (the consent form must be signed by the subject prior to any study-specific procedures), and evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study;
* Willingness and ability to comply with study procedures and follow-up examination.
* Adequate organ function as evidenced by the following peripheral blood counts or serum chemistry values within 28 days before randomization:

  1. Hemoglobin greater than or equal to 9 g/dL
  2. Neutrophil count (ANC) greater than or equal to 1,500/microL
  3. Platelet count greater than or equal to 100,000/microL
  4. Serum creatinine less than or equal to 1.5 mg/dL (less than or equal to 132.6 micromol/L) and creatinine clearance greater than or equal to 60 ml/min
  5. Creatine phosphokinase (CPK) less than or equal to 2x upper limit of normal (ULN)
  6. Hepatic function variables:

     1. Total bilirubin ≤ 1.5x ULN
     2. Total alkaline phosphatase (ALP) ≤ 1.5x ULN, or if > 1.5x ULN, then ALP liver fraction or 5' nucleotidase must be ≤1x ULN
     3. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) must be ≤ 2.5x ULN

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease.
* Subjects with a history of hypersensitivity to edaravone or any of the inactive ingredients of the formulation (such as sulfite and sodium bisulfite).
* Subjects with PR >240 msec, QRS =120 msec, or QTcF >450 msec for male & QTcF >470 msec for female on the screening or Day -1 ECG, or any clinically significant electrocardiographic abnormality in the opinion of the investigator.
* Male subjects with partners currently pregnant; male subjects able to father children who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study and for at least 3 months after the last dose of investigational product.
* Female subjects currently pregnant or lactating; female subjects able to bear children or of child bearing potential who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study and for at least 3 months after the last dose of investigational product.
* Subjects whose urine drug/alcohol screening was positive at the time of screening and/or on Day-1.
* Subjects having difficulty in swallowing pills/tablets.
* Subjects smoking > 5 cigarettes per day within 3 months prior to the screening visit.
* Subjects unwilling or unable to comply with the Lifestyle Guidelines described in the protocol.
* Subjects who are investigational site staff members directly involved in the conduct of the studies and their family members, site staff members otherwise supervised by the Investigator, or subjects who are the sponsors' employees directly involved in the conduct of the studies.
* Evidence of any severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this trial.
* Subjects who have participated in another clinical trial less than 3 months before or donated his/her blood in a quantity greater than 200 milliliters (mL) within 1 month of the screening period of this clinical trial.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2020-04-24 (Actual); Primary Completion 2020-12-17 (Actual); Study Completion 2021-01-08 (Actual)

PRIMARY OUTCOMES:
Adverse events | until the last follow-up visit, up to 4 weeks
  Frequencies (number and percentage) of subjects with one or more AEs
change in hemoglobin (g/L) | up to 6 days post each dose
  measured by hematology test
change in hematocrit (ratio) | up to 6 days post each dose
  measured by hematology test
change in red blood cell count (cells x 10^12/L) | up to 6 days post each dose
  measured by hematology test
change in white blood cell (WBC) count (cells x 10^9/L) | up to 6 days post each dose
  measured by hematology test
change in platelet count (cells x 10^9/L) | up to 6 days post each dose
  measured by hematology test
change in total neutrophils count (cells x 10^9/L) | up to 6 days post each dose
  measured by hematology test
change in lymphocytes count (cells x 10^9/L) | up to 6 days post each dose
  measured by hematology test
change in monocytes count (cells x 10^9/L) | up to 6 days post each dose
  measured by hematology test
change in eosinophils count (cells x 10^9/L) | up to 6 days post each dose
  measured by hematology test
change in basophils count (cells x 10^9/L) | up to 6 days post each dose
  measured by hematology test
change in serum sodium (mmol/L) | up to 6 days post each dose
  measured by serum chemistry
change in serum potassium (mmol/L) | up to 6 days post each dose
  measured by serum chemistry
change in serum chloride (mmol/L) | up to 6 days post each dose
  measured by serum chemistry
change in serum calcium (mmol/L) | up to 6 days post each dose
  measured by serum chemistry
change in serum glucose (mmol/L) | up to 6 days post each dose
  measured by serum chemistry
change in serum urea (mmol/L) | up to 6 days post each dose
  measured by serum chemistry
change in serum creatinine (umol/L) | up to 6 days post each dose
  measured by serum chemistry
change in serum total bilirubin (umol/L) | up to 6 days post each dose
  measured by serum chemistry
change in aspartate aminotransferase (AST) (U/L) | up to 6 days post each dose
  measured by serum chemistry
change in alanine aminotransferase (ALT) (U/L) | up to 6 days post each dose
  measured by serum chemistry
change in alkaline phosphatase (ALP) (U/L) | up to 6 days post each dose
  measured by serum chemistry
change in serum creatine kinase (CK) (U/L) | up to 6 days post each dose
  measured by serum chemistry
change in serum albumin (g/L) | up to 6 days post each dose
  measured by serum chemistry
change in serum phosphate (mmol/L) | up to 6 days post each dose
  measured by serum chemistry
change in serum lipase (U/L) | up to 6 days post each dose
  measured by serum chemistry
change in serum total protein (g/L) | up to 6 days post each dose
  measured by serum chemistry
change in urine pH | up to 6 days post each dose
  measured by urinalysis
change in urine specific gravity | up to 6 days post each dose
  measured by urinalysis
change in urine glucose | up to 6 days post each dose
  measured by urinalysis
change in urine protein | up to 6 days post each dose
  measured by urinalysis
change in urine ketones | up to 6 days post each dose
  measured by urinalysis
change in urine blood | up to 6 days post each dose
  measured by urinalysis
change in urine casts | up to 6 days post each dose
  measured by microscopic analysis, if any abnormalities in urinalysis are detected
change in urine crystals | up to 6 days post each dose
  measured by microscopic analysis, if any abnormalities in urinalysis are detected
change in urine epithelial cells | up to 6 days post each dose
  measured by microscopic analysis, if any abnormalities in urinalysis are detected
change in urine bacteria (cfu/L) | up to 6 days post each dose
  measured by microscopic analysis, if any abnormalities in urinalysis are detected
change in urine red blood cells (Cells x 10^9/L) | up to 6 days post each dose
  measured by microscopic analysis, if any abnormalities in urinalysis are detected
change in urine white blood cells (Cells x 10^9/L) | up to 6 days post each dose
  measured by microscopic analysis, if any abnormalities in urinalysis are detected
change in systolic blood pressure (mmHg) | up to 6 days post each dose
change in diastolic blood pressure (mmHg) | up to 6 days post each dose
change in pulse rate (bpm) | up to 6 days post each dose
change in body temperature (celsius) | up to 6 days post each dose
Change in QT intervals (msec) | up to 6 days post each dose
  Measured using a 12 Lead Electrocardiogram
Change in RR intervals (msec) | up to 6 days post each dose
  Measured using a 12 Lead Electrocardiogram
Change in PR intervals (msec) | up to 6 days post each dose
  Measured using a 12 Lead Electrocardiogram
Change in QRS duration (msec) | up to 6 days post each dose
  Measured using a 12 Lead Electrocardiogram
Change in corrected QTcF (msec) | up to 6 days post each dose
  Calculated using measurements by a 12 Lead Electrocardiogram
clinically significant abnormality in brief physical examinations | up to 6 days post each dose
  clinically significant abnormality in skin, lungs, cardiovascular system, and abdomen (spleen and liver)

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | up to 24 hours post each dose
Time of maximum plasma concentration (Tmax) | up to 24 hours post each dose
Area under the plasma concentration-time curve from time-zero extrapolated to infinite time (AUC0-inf) | up to 24 hours post each dose
Area under the plasma concentration-time curve from time-zero to the time of the last measurable concentration (AUC0-last) | up to 24 hours post each dose
The ratio of area under the plasma concentration-time curve from time-zero to the time of the last measurable concentration (AUC0-last) extrapolated to AUC0-inf over AUC0-inf (% AUCex) | up to 24 hours post each dose
Apparent volume of distribution (Vd/F) | up to 24 hours post each dose
Terminal half-life(T1/2) | up to 24 hours post each dose
Apparent oral clearance (CL/F) | up to 24 hours post each dose
Mean retention time (MRT) | up to 24 hours post each dose
Lambda z - the reciprocal of elimination rate constant (λz) | up to 24 hours post each dose
Fabs-bioavailability value (Fabs) | up to 24 hours post each dose

CONTACTS AND LOCATIONS:
Overall Officials: Sepehr Shakib, MD, Principal Investigator — Royal Adelaide Hospital
Locations (1):
- CMAX Clinical Research Pty Ltd, Adelaide, South Australia, Australia